CLINICAL TRIAL: NCT06407310
Title: Phase II Open-label, Single-arm Trial of Neoadjuvant Pembrolizumab With Carboplatin and Paclitaxel in Triple-negative Breast Cancer
Brief Title: Neoadjuvant Pembrolizumab, Carboplatin and Paclitaxel in Triple-negative Breast Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, Yasmin Leshem, Senior Medical Oncologist, Tel Aviv Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0617-22 TLV
Record Dates: First submitted 2024-03-04; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Triple Negative Breast Cancer
Keywords: Immunotherapy; Pembrolizumab; Breast cancer; Triple-negative breast cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Breast Neoplasms | interventions — pembrolizumab; Carboplatin; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Masking Description: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- neoadjuvant pembrolizumab with carboplatin and paclitaxel in triple-negative breast cancer (Experimental): 6 cycles of Pembrolizumab (Keytruda) at a dose of 200 mg given every 3 weeks for 6 cycles. The first cycle of pembrolizumab is given as a lead-in without carboplatin and paclitaxel.
  Carboplatin area under the curve (AUC) 1.5 and Paclitaxel 80 mg/m2, starting with the second pembrolizumab cycle, will be given weekly for 12 weeks.
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Paclitaxel

INTERVENTIONS:
Drug: Pembrolizumab — I.V Pembrolizumab (keytruda) 200 mg every 3 weeks for 6 cycles
Drug: Carboplatin — I.V Carboplatin at AUC 1.5 weekly for a total of 12 weeks.
Drug: Paclitaxel — I.V Paclitaxel at 80 mg/m2 weekly for a total of 12 weeks.

SUMMARY:
This is a phase II, single-centered, open-label, single-armed study in patients with early triple-negative breast cancer that will evaluate the pathological complete response (pCR) rate of a non-anthracycline-based chemo-immunotherapy regimen. The trial includes a lead-in cycle of pembrolizumab, then a combination of paclitaxel, carboplatin, and pembrolizumab in the neoadjuvant setting.

DETAILED DESCRIPTION:
The cure rate of stage I and II triple-negative breast cancer treated with anthracycline-based chemotherapy is high but comes at the price of substantial toxicity. This is a phase II, single-centered, open-label, single-armed study in patients with early triple-negative breast cancer that will evaluate the pathological complete response (pCR) rate and immune effects of a non-anthracycline-based chemo-immunotherapy regimen. The trial includes a lead-in cycle of pembrolizumab, then a combination of paclitaxel, carboplatin, and pembrolizumab in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female participants who are at least 18 years of age on the day of signing informed consent with a histologically confirmed diagnosis of stage I or II TNBC.
2. Tumor size of above 1 cm.
3. The patient is willing to provide tissue from newly obtained core biopsies.
4. Male participants:

   A male participant must agree to use contraception as detailed in Appendix 3 of this protocol during the treatment period and for at least 200 days after the last dose of study treatment and refrain from donating sperm during this period.
5. Female participants:

   A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:
   1. Not a woman of childbearing potential (WOCBP). OR
   2. A WOCBP who agrees to follow the contraceptive during the treatment period and for at least 180 days after the last dose of chemotherapy.
6. The participant (or legally acceptable representative if applicable) provides written informed consent for the trial.
7. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1. Evaluation of ECOG is to be performed within 7 days before the first dose of study intervention.
8. Have adequate organ function as defined in the following table (Table 4). Specimens must be collected within 10 days before the start of the study intervention.
9. Criteria for known Hepatitis B and C positive subjects

Hepatitis B (HBV) and C (HCV) screening tests are not required unless:

* Known history of HBV or HCV infection
* As mandated by the local health authority

10.1 Hepatitis B positive subjects:

* Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have an undetectable HBV viral load before randomization.
* Participants should remain on anti-viral therapy throughout the study intervention and follow local guidelines for HBV anti-viral therapy post-completion of the study intervention.

10.2 Participants with a history of HCV infection are eligible if the HCV viral load is undetectable at screening.

• Participants must have completed curative anti-viral therapy at least 4 weeks before randomization.

Exclusion Criteria:

1. A WOCBP who has a positive urine pregnancy test within 72 hours prior of the first treatment dose (. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
2. Has received prior therapy with an anti-Programmed cell death-ligand-1 (PD-L1), anti-PD-1, or anti-PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, cytotoxic T-lymphocyte associated protein 4 (CTLA-4), OX 40, CD137).
3. Has received prior systemic anti-cancer therapy, including investigational agents, within 24 months of screening.
4. Has received prior radiotherapy within 24 months of screening.
5. Has received a live vaccine or live-attenuated vaccine within 30 days before the first dose of study intervention. Administration of killed vaccines is allowed.

   Note: please refer to Section 5.5.2 for information on coronavirus disease 2019 (COVID-19) vaccines
6. Has received an investigational agent or has used an investigational device within 4 weeks before study intervention administration.
7. Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of the study drug.
8. Known additional malignancy that is progressing or has required active treatment within the past 3 years. Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.
9. Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years except for replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid).
11. Has a history of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
12. Has an active infection requiring systemic therapy.
13. Has a known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authorities.
14. Concurrent active Hepatitis B (defined as HBsAg positive and/or detectable HBV DNA) and Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA) infection.

    Note: Hepatitis B and C screening tests are not required unless:
    * Known history of HBV and HCV infection
    * As mandated by the local health authority
15. Has not adequately recovered from major surgery or has ongoing surgical complications.
16. Has a history or current evidence of any condition, therapy, laboratory abnormality, or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
17. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment or 180 after the last dose of chemotherapy.
19. Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate (pCR= ypT0/Tis ypN0) | 3 years
  The number of patients with pathological complete response (pCR) out of the total number of trial participants using a definition of ypT0/Tis ypN0 after treatment with neoadjuvant pembrolizumab, paclitaxel and carboplatin (PCb).
Molecular dynamics of cells in the tumor microenvironment (TME) | 3 years
  The molecular state of cells in the TME will be measured at a single-cell level using single-cell RNA sequencing (scRNA-seq) before and after one dose of pembrolizumab.

SECONDARY OUTCOMES:
3-year overall survival (OS) rate | 5 years
  The number of patients that are alive three years after entering the trial out of the total number of trial participants.
3-year event-free survival (EFS) rate | 5 years
  The number of patients without disease recurrence three years after entering the trial out of the total number of trial participants.

IPD SHARING:
Plan to Share IPD: No